CLINICAL TRIAL: NCT00954421
Title: Use of Two DBS Electrodes to Treat Post-Traumatic Tremor
Brief Title: Use of Two Deep Brain Stimulation (DBS) Electrodes to Treat Post-Traumatic Tremor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 461-2006; K23NS052557 (NIH)
Record Dates: First submitted 2009-07-27; First posted 2009-08-07 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Deep Brain Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Deep Brain Stimulation (Experimental): Multiple Sclerosis Tremor treated with VIM and VO Deep Brain Stimulation
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Use of two ipsilateral thalamic Deep Brain Stimulation electrodes (one at the ventralis intermedius nucleus/ventralis oralis posterior nucleus border or VIM and one at the ventralis oralis anterior nucleus/ventralis oralis posterior nucleus border or VO) for treatment of disabling and medication refractory tremor secondary to head trauma or multiple sclerosis.

SUMMARY:
The purpose of this research study is to:

1. Determine whether deep brain stimulation (DBS) with two leads (very thin coiled wires) placed unilaterally (on one side of the brain) is beneficial to patients with multiple sclerosis (MS) tremor.
2. Compare the two different locations of the DBS lead placement in effectiveness for treatment of muscle tremors that do not respond to treatment with medication caused by multiple sclerosis.
3. Evaluate any side effects that may result from the two DBS leads.

DETAILED DESCRIPTION:
Surgical treatment of disabling multiple sclerosis (MS) tremor that does not respond to medication has proven difficult. To date, there have been no prospective blinded studies to evaluate efficacy of surgical treatments for these tremors. Based on prior data, this study will examine the use of 2 DBS electrodes on the same side of the brain in the thalamus region (one at an area referred to as the "ventralis intermedius nucleus/ventralis oralis posterior nucleus border," or "VIM," and one at a region called the "ventralis oralis anterior nucleus/ventralis oralis posterior nucleus border," or "VO") for treatment of MS tremor. This study will test the effectiveness of VIM combined with, and independent of, VO DBS, and characterize safety, benefits and side effects of this procedure for treatment of MS-related tremors.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have an unequivocal diagnosis of Multiple Sclerosis (MS) resulting in disabling tremor as indicated by a score of at least 3 on the Tremor Rating Scale (TRS) baseline global assessments by the examiner and the patient.
* The patient must have a history of an unsatisfactory response to medical management. Any patient will need to have tried and failed at least one drug from at least three of the four following medication classes: anticholinergics, muscle relaxants, benzodiazepines, and beta blockers. Alternatively, a patient may also qualify if tremor-suppressing medications are contraindicated due to a coexisting medical condition or drug allergy.
* The MS patient must have disabling and medically refractory unilateral or bilateral upper extremity tremor. Patients with associated ipsilateral lower extremity tremor are not excluded.
* The tremor must meet the following specific diagnostic criteria:

  * The tremor must be predominantly postural or action (versus resting) and have a rhythmic and/or ballistic characteristic.
  * The tremor may not have features that indicate a significant cerebellar etiology (i.e., non-prominent ataxia, dysdiadokokinesia, dysmetria).
  * The tremor must have been present and either stable or progressing for greater than one year.
  * The tremor must be disabling. Disabling is defined as significant impairment of the normal functions of daily life as indicated by a score of at least 5 on the Clinical Global Impression (CGI)-Severity scale.

Exclusion Criteria:

* Significant medical disease that would excessively increase risk of peri-operative complications (significant cardiac or pulmonary disease, uncontrolled hypertension, inadequately treated major depression).
* More than mild non-tremor cerebellar dysfunction (ataxia, dysmetria, dysdiadokokinesia).
* Evidence of secondary/atypical movement disorder as suggested by presence of the following:

  * history of stroke(s)
  * exposure to toxins or neuroleptics
  * history of encephalitis
  * neurological signs of upper motor neuron disease, supranuclear gaze palsy, or significant orthostatic hypotension
* MRI with significant evidence of severe brain atrophy or other prohibitive abnormalities (absence of thalamic target for Deep Brain Stimulation (DBS), lacunar infarcts, or iron deposits in the putamen).
* Cognitive dysfunction as evidenced by a score of less than 120 on the Mattis Dementia Rating Scale (MDRS) Such patients will be excluded because significant dementia places the patient at high risk for surgery-induced deterioration of cognitive function, and such patients might have limited ability to accurately assess the impact of DBS.
* Major psychiatric disorder on the Structured Clinical Interview (SCID-IV) for the Diagnostic and Statistical Manual Version 4 (DSM-IV). 45 Patients with Major Depression within 3 months of entry into the study will be excluded. High rates of psychiatric co-morbidity can complicate any neurosurgical study. While the cleanest study would exclude patients with psycho-pathology, we do not believe this is realistic or practical, given the majority of patients with advanced movement disorders will suffer from some degree of anxiety or depression. We will screen patients for psychiatric disorders, treat disorders prior to DBS and admit patients who are psychiatrically stable for at least 3 months prior to entry (without active psychiatric diagnosis by SCID criteria).
* Patients with any implanted device that precludes magnetic resonance imaging (MRI) will be excluded from this study. Examples of such devices include cochlear implants, spinal cord stimulators, many cardiac pacemakers, and some older aneurysm clips
* Patients who have a known need for future MRIs or diathermy treatments will be excluded from this study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-11; Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Foote, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Oliveria SF, Rodriguez RL, Bowers D, Kantor D, Hilliard JD, Monari EH, Scott BM, Okun MS, Foote KD. Safety and efficacy of dual-lead thalamic deep brain stimulation for patients with treatment-refractory multiple sclerosis tremor: a single-centre, randomised, single-blind, pilot trial. Lancet Neurol. 2017 Sep;16(9):691-700. doi: 10.1016/S1474-4422(17)30166-7. Epub 2017 Jun 20. PMID 28642125

RESULTS

PARTICIPANT FLOW:
Groups:
- Multiple Sclerosis Tremor On VIM and VO: Multiple Sclerosis Tremor On VIM and VO Deep Brain Stimulation
  Deep Brain Stimulation: Use of two ipsilateral thalamic Deep Brain Stimulation electrodes (one at the ventralis intermedius nucleus/ventralis oralis posterior nucleus border or VIM and one at the ventralis oralis anterior nucleus/ventralis oralis posterior nucleus border or VO) for treatment of disabling and medication refractory tremor secondary to head trauma or multiple sclerosis.
Period: Screening
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 16
Completed | 13
Not Completed | 3
Not completed — screen failures | 3
Period: Baseline
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 13
Completed | 13
Not Completed | 0
Period: 6 Months of DBS
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 13
Completed | 12
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: VIM=ON VO=ON at 6 Months
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 12 (This is the point of evaluation: Order of assessment was random for periods 4-7)
Completed | 12
Not Completed | 0
Period: VIM=OFF VO=OFF at 6 Months
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 12
Completed | 12
Not Completed | 0
Period: VIM=OFF VO=ON at 6 Months
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 12
Completed | 12
Not Completed | 0
Period: VIM=ON VO=OFF at 6 Months
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All eligible subjects were enrolled and the intent was to treat for six months on dual lead deep brain stimulation in the VIM and VO regions.
Arm/Group | All Subjects
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.54 (15.03)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 13
Baseline Total Fain-Tolosa-Marin Tremor Rating Scale (TRS) [Mean (Standard Deviation); unit: units on a scale] — Tremor was evaluated using the Fain-Tolosa-Marin Tremor Rating Scale (TRS). Score was obtained by summing all 21 items, each of which assessed tremor on a scale of 0-4. Because some of the 21 items contained more than one subsection, total maximum score was 144, and minimum score was 0. Higher scores represent worse tremor.
  units on a scale | 56.2 (9.4)

OUTCOME MEASURES:

1. Primary Outcome: Fain-Tolosa-Marin Tremor Rating Scale (TRS) Change Score for Both VIM and VO ON (Baseline Minus 6 Months Post-implant)
Description: Tremor was evaluated using the Fain-Tolosa-Marin Tremor Rating Scale (TRS). Score was obtained by summing all 21 items, each of which assessed tremor on a scale of 0-4. Because some of the 21 items contained more than one subsection, total maximum score was 144, and minimum score was 0. Higher scores represent worse tremor.
  Both VIM and VO stimulators will be turned ON and TRS score at 6 months will be compared to pre-implant (baseline).
Time Frame: Change from Baseline to Six Months
Population: All Subjects completing Period 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Number analyzed (Participants) | 12
units on a scale | -17.6 (19.4)
Statistical Analysis 1: Comparison: Multiple Sclerosis Tremor On VIM and VO; The null hypothesis is that the mean change in Tremor Rating Scale score from baseline to six months post-implant (with VIM and VO stimulators turned ON) will be zero; Test type: Superiority or Other; p = .026, two-sided sign-rank test; Mean Difference (Net) = -17.6, 95% CI 2-sided [-30.61 to -4.65], Standard Deviation 19.4 — p-value assessed via sign-rank test (pre-planned method)

2. Secondary Outcome: Fain-Tolosa-Marin Tremor Rating Scale (TRS) Change Score for Either VIM or VO On, and for Both VIM and VO Off (Baseline Minus 6 Months Post-implant)
Description: Tremor was evaluated using the Fain-Tolosa-Marin Tremor Rating Scale (TRS). Score was obtained by summing all 21 items, each of which assessed tremor on a scale of 0-4. Because some of the 21 items contained more than one subsection, total maximum score was 144, and minimum score was 0. Higher scores represent worse tremor.
  Both VIM and VO stimulators will be turned ON and TRS score at 6 months will be compared to pre-implant (baseline).
  Either VO or VIM stimulator will be turned on (as opposed to both stimulators, as in outcome measure 1), and change in Tremor Rating Scale scores will be compared. The effects of each individual stimulator will also be compared to both being turned on.
Time Frame: Baseline to Six Months
Population: Patients completing 6 months were tested for VIM and VO both on vs. both off. Score is TRS scale with both off minus both on. Positive value favors DBS.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TRS Scale Both Off vs Both on at 6 Months: Multiple Sclerosis Tremor On VIM and VO Deep Brain Stimulation Periods 4 vs. 5(Both OFF- Both On) at 6 months.
  Deep Brain Stimulation: Use of two ipsilateral thalamic Deep Brain Stimulation electrodes (one at the ventralis intermedius nucleus/ventralis oralis posterior nucleus border or VIM and one at the ventralis oralis anterior nucleus/ventralis oralis posterior nucleus border or VO) for treatment of disabling and medication refractory tremor secondary to head trauma or multiple sclerosis.
- TRS Scale Vo Only on vs. Vim Only on at 6 Months: Multiple Sclerosis Tremor On VIM and VO Deep Brain Stimulation Periods 4 vs. 5(Vo only on -VM only on at 6 months.
  Deep Brain Stimulation: Use of two ipsilateral thalamic Deep Brain Stimulation electrodes (one at the ventralis intermedius nucleus/ventralis oralis posterior nucleus border or VIM and one at the ventralis oralis anterior nucleus/ventralis oralis posterior nucleus border or VO) for treatment of disabling and medication refractory tremor secondary to head trauma or multiple sclerosis.
Arm/Group | TRS Scale Both Off vs Both on at 6 Months | TRS Scale Vo Only on vs. Vim Only on at 6 Months
Number analyzed (Participants) | 12 | 11
units on a scale | 8.4 (9.1) | 0.73 (8.49)
Statistical Analysis 1: Comparison: TRS Scale Both Off vs Both on at 6 Months; The null hypothesis is that difference in change in Tremor Rating Scale (TRS) score from baseline to 6 months when both stimulators are on (VIM and VO), versus when both stimulators are off, will be zero (i.e., that there will be no difference in effect between having both stimulators on versus both stimulators off); Test type: Superiority or Other; p = 0.011, Sign-Rank test — Sign rank test was pre-planned for P-value; Mean Difference (Net) = 8.4, 95% CI 2-sided [2.2 to 14.5], Standard Deviation 9.1 — p-value assessed using sign rank test
Statistical Analysis 2: Comparison: TRS Scale Vo Only on vs. Vim Only on at 6 Months; The null hypothesis is that difference in change in Tremor Rating Scale (TRS) score from baseline to 6 months when VO is on and VIM is off, versus when VIM is on and VO is off, will be zero (i.e., that there will be no difference in effect between having exclusively VIM versus VO on); Test type: Superiority or Other; p = .68, two-sided sign rank test; two sided sign rank test as pre-planned; Mean Difference (Net) = .73, 95% CI [-4.96 to 6.42], Standard Deviation 8.49

ADVERSE EVENTS:
Time Frame: Baseline, 6 months, 24 months
Arm/Group | Multiple Sclerosis Tremor On VIM and VO
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Sclerosis Tremor On VIM and VO (N=13)
Superficial Wound Infection (Infections and infestations) | 1 (1)
Infection at site of IPG (pulse generator for DBS implant) (Infections and infestations) | 1 (1)
Death (Injury, poisoning and procedural complications) | 1 (1) — drowning due to accident (related to her multiple sclerosis)
Change in mental status (Psychiatric disorders) | 2 (2)
Exacerbation of Multple Sclerosis symptoms (Nervous system disorders) | 1 (3) — affecting facial never numbness (1 case), progressive weakening (2 cases)
Right fractured femur (Injury, poisoning and procedural complications) | 1 (1)
Complications with device hardware (Surgical and medical procedures) | 2 (2) — fractured DBS cables (1 case), erosion over hardware (1 case)
Implantation of tunneled intrathecal catheter and subcutaneous implantation of a programmable pump (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Multiple Sclerosis Tremor On VIM and VO (N=13)
Clostridium Difficile Infection (Infections and infestations) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Gastrointestinal discomfort (Gastrointestinal disorders) | 3 (6) — diarrhea (1 case), nausea (1 case), vomiting (1 case), constipation (2 cases)
speech difficulty (General disorders) | 4 (6) — slurred speech (3 cases), slower speech (2 cases), stuttering speech (1 case)
swallowing difficulty (General disorders) | 1 (1)
lightheadedness (General disorders) | 1 (2)
facial numbness (Nervous system disorders) | 1 (1)
trigeminal neuralgia (Nervous system disorders) | 1 (1)
weakness (Musculoskeletal and connective tissue disorders) | 3 (5)
decreased mobility (Musculoskeletal and connective tissue disorders) | 2 (5)
worsened balance (General disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 3 (5)
worsening of nasal allergies (Immune system disorders) | 1 (1)
laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
headache (General disorders) | 6 (8)
pain behind left ear (General disorders) | 1 (1)
pain under left eye (General disorders) | 1 (1)
neck pain (General disorders) | 1 (1)
back pain (General disorders) | 1 (1)
lower breast pain (General disorders) | 1 (1)
internal capsule pulling (General disorders) | 1 (1)
pain on left side of head (General disorders) | 1 (1)
crying (Psychiatric disorders) | 3 (3)
irritability (Psychiatric disorders) | 1 (1)
scalp tenderness (Injury, poisoning and procedural complications) | 1 (1)
head pain at crania cap (Injury, poisoning and procedural complications) | 1 (1)
pinching at site of pulse generator (Injury, poisoning and procedural complications) | 2 (2)
Twiddler syndrome (Nervous system disorders) | 2 (2)
scar tissue formation at site of DBS (Injury, poisoning and procedural complications) | 1 (1)
irritation at site of pulse generator (Injury, poisoning and procedural complications) | 3 (3)
urinary tract infection (Infections and infestations) | 2 (3)
eczema (General disorders) | 1 (1)
intra-operative seizure (Nervous system disorders) | 1 (1)
fatigue (Psychiatric disorders) | 4 (5)
eyelid fluttering (Eye disorders) | 1 (2)
tremor in bottom lip (Nervous system disorders) | 1 (1)
tremor in abdomen (Psychiatric disorders) | 1 (1)
insomnia (Psychiatric disorders) | 2 (2)
nocturnal myoclonus of lower extremities (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes